CLINICAL TRIAL: NCT03108066
Title: An Open Label Phase 2 Study to Evaluate PT2385 for the Treatment of Von Hippel-Lindau Disease-Associated Clear Cell Renal Cell Carcinoma
Brief Title: MK-3795 (PT2385) for the Treatment of Von Hippel-Lindau Disease-Associated Clear Cell Renal Cell Carcinoma (MK-3795-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peloton Therapeutics, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3795-003; PT2385-202 (Other: Peloton Study ID); MK-3795-003 (Other: MSD)
Record Dates: First submitted 2017-03-28; First posted 2017-04-11 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: VHL Gene Mutation; VHL; VHL Syndrome; VHL Gene Inactivation; Von Hippel; Von Hippel-Lindau Disease; Von Hippel's Disease; Von Hippel-Lindau Syndrome, Modifiers of; Clear Cell Renal Cell Carcinoma; Clear Cell RCC; ccRCC
MeSH Terms: conditions — von Hippel-Lindau Disease; Carcinoma, Renal Cell | interventions — PT2385

STUDY DESIGN:
Intervention Model Description: This is an open-label Phase 2 study that will be conducted with a 2-stage design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-3795 (Experimental): Participants receive 800 mg MK-3795 orally twice daily. Participants may continue to receive MK-3795 in the absence of unacceptable treatment related toxicity or unequivocal disease progression.
  Interventions: Drug: MK-3795

INTERVENTIONS:
Drug: MK-3795 — 800 mg twice daily (four 200 mg oral tablets twice daily)
  Other Names: PT2385, PT-2385

SUMMARY:
The primary objective of this study is to assess the overall response rate (ORR) of von Hippel-Lindau (VHL) disease-associated clear cell renal cell carcinoma (ccRCC) tumors in VHL participants treated with MK-3795.

DETAILED DESCRIPTION:
This open-label Phase 2 study will evaluate the efficacy, safety, PK, and PD of MK-3795 in participants with VHL disease who have at least 1 measurable VHL disease-associated ccRCC tumor (as defined by RECIST 1.1). MK-3795 will be administered orally and treatment will be continuous. Changes in VHL disease-associated non-ccRCC tumors will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Has at least 1 measurable ccRCC tumor and no solid ccRCC tumor greater than 3.0 cm, based on radiologic diagnosis (histologic diagnosis not required); may have VHL disease-associated lesions in other organ systems
* Has a diagnosis of von Hippel Lindau disease, based on a germline VHL alteration

Exclusion Criteria:

* Has had prior radiotherapy or systemic anti cancer therapy for ccRCC (includes anti-vascular endothelial growth factor (VEGF) therapy or any systemic investigational anti cancer agent)
* Has a prior or concomitant non-VHL disease-associated invasive malignancy with the exception of adequately treated basal or squamous cell carcinoma of the skin, cervical carcinoma in situ or any other malignancy from which the participant has remained disease free for more than 2 years
* Has any history of metastatic disease
* Has had radiotherapy to any non-ccRCC site within 4 weeks prior to entering the study or has not recovered from adverse events (AE)
* Has had any surgical procedure for VHL disease or any major surgical procedure completed within 4 weeks prior to entering the study or has any surgical lesions from recent major surgical procedures that are not well healed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Larcher A, Rowe I, Belladelli F, Fallara G, Raggi D, Necchi A, Montorsi F, Capitanio U, Salonia A; OSR VHL Program. Von Hippel-Lindau disease-associated renal cell carcinoma: a call to action. Curr Opin Urol. 2022 Jan 1;32(1):31-39. doi: 10.1097/MOU.0000000000000950. PMID 34783716
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-3795: Participants received 800 mg MK-3795 orally twice daily. Participants continued to receive MK-3795 in the absence of unacceptable treatment related toxicity or unequivocal disease progression.
Period: Overall Study
Arm/Group | MK-3795
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MK-3795
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) in VHL Disease-Associated ccRCC Tumors
Description: ORR was defined as the percentage of participants in the analysis population who have a best confirmed response of Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). ORR was assessed by independent review committee (ICR) for the primary analysis.
Time Frame: Up to approximately 76 months
Population: The analysis population consisted of all allocated participants who received at least one dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-3795
Number analyzed (Participants) | 4
Percentage of Participants | 0.0 [0.0 to 60.2]

2. Secondary Outcome: Progression-free Survival (PFS) in VHL Disease-Associated ccRCC Tumors
Description: PFS was defined as the interval from the start of study treatment to the first documented Progressive Disease (PD) or death from any cause, whichever occurs first. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD.
Time Frame: Up to approximately 76 months
Population: The analysis population consisted of all allocated participants who received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MK-3795
Number analyzed (Participants) | 4
Months | NA [NA to NA] — NA = Median, upper limit, and lower limit not reached at time of data cut-off due to insufficient number of participants with an event.

3. Secondary Outcome: Duration of Response (DOR) in VHL Disease-Associated ccRCC Tumors
Description: DOR was defined as the interval from the first documented evidence of a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 until PD or death due to any cause, whichever occurs first, in participants demonstrating a best confirmed response of CR or PR. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD.
Time Frame: Up to approximately 76 months
Population: The analysis population consisted of all allocated participants who received at least one dose of study intervention and experienced CR or PR. No participants experienced CR or PR and DOR was not analyzed.
Arm/Group | MK-3795
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Response (TTR) in VHL Disease-Associated ccRCC Tumors
Description: TTR was defined as the interval from the start of study treatment to the first documentation of a response per RECIST 1.1, and calculated for participants with a best confirmed response of CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions).
Time Frame: Up to approximately 76 months
Population: The analysis population consisted of all allocated participants who received at least one dose of study intervention and experienced CR or PR. No participants experienced CR or PR and TTR was not analyzed.
Arm/Group | MK-3795
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Response Rate (ORR) in VHL Disease-Associated Non-ccRCC Tumors
Description: ORR was defined as the percentage of participants in the analysis population who have a best confirmed response of Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).
Time Frame: Up to approximately 76 months
Population: There were no reported non-ccRCC tumors in allocated participants, therefore no analysis was performed.
Arm/Group | MK-3795
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression-free Survival (PFS) in VHL Disease-Associated Non-ccRCC Tumors
Description: PFS was defined as the interval from the start of study treatment to the first documented PD or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD.
Time Frame: Up to approximately 76 months
Population: There were no reported non-ccRCC tumors in allocated participants, therefore no analysis was performed.
Arm/Group | MK-3795
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of Response (DOR) in VHL Disease-Associated Non-ccRCC Tumors
Description: DOR was defined as the interval from the first documented evidence of a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 until Progressive Disease (PD) or death due to any cause, whichever occurs first, in participants demonstrating a best confirmed response of CR or PR. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD.
Time Frame: Up to approximately 76 months
Population: There were no reported non-ccRCC tumors in allocated participants, therefore no analysis was performed.
Arm/Group | MK-3795
Number analyzed (Participants) | 0

8. Secondary Outcome: Time to Response (TTR) in VHL Disease-Associated Non-ccRCC Tumors
Description: as for outcome 4
Time Frame: Up to approximately 76 months
Population: There were no reported non-ccRCC tumors in allocated participants, therefore no analysis was performed.
Arm/Group | MK-3795
Number analyzed (Participants) | 0

9. Secondary Outcome: MK-3795 Plasma Concentration
Description: Blood samples for the determination of MK-3795 concentration were collected at pre-specified timepoints before and after administration of study intervention.
Time Frame: Week 1: pre-dose and 6 hours post-dose, Week 3, 5, 9, 13, and 17: pre-dose
Population: The analysis population consisted of all allocated participants who received at least one dose of study intervention and had available MK-3475 plasma concentration data at the specified timepoints. No participants had available MK-3475 plasma concentration data at Week 17.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MK-3795
Number analyzed (Participants) | 4
ng/mL
  Week 1 Pre-dose | NA (NA) — NA means not calculable as MK-3795 could not be detected.
  Week 1 6 Hours Post-dose | 583 (104.6)
  Week 3 Pre-dose: number analyzed (Participants) | 2
  Week 3 Pre-dose | 1750 (76.8)
  Week 5 Pre-dose: number analyzed (Participants) | 2
  Week 5 Pre-dose | 1480 (93.5)
  Week 9 Pre-dose: number analyzed (Participants) | 1
  Week 9 Pre-dose | 2550 (NA) — Geometric Coefficient of Variation could not be calculated if the number of participants analyzed was less than 2.
  Week 13 Pre-dose: number analyzed (Participants) | 1
  Week 13 Pre-dose | 3150 (NA) — Geometric Coefficient of Variation could not be calculated if the number of participants analyzed was less than 2.
  Week 17 Pre-dose: number analyzed (Participants) | 0

10. Secondary Outcome: MK-3795 Metabolite Plasma Concentration
Description: Blood samples for the determination of MK-3795 metabolite concentration were collected at pre-specified timepoints before and after administration of study intervention.
Time Frame: Week 1: pre-dose and 6 hours post-dose, Week 3, 5, 9, 13, and 17: pre-dose
Population: The analysis population consisted of all allocated participants who received at least one dose of study intervention and had available MK-3475 metabolite plasma concentration data at the specified timepoints. No participants had available MK-3475 metabolite plasma concentration data at Week 17.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MK-3795
Number analyzed (Participants) | 4
ng/mL
  Week 1 Pre-dose | NA (NA) — NA means not calculable as MK-3795 metabolite could not be detected.
  Week 1 6 Hours Post-dose | 2790 (95.5)
  Week 3 Pre-dose: number analyzed (Participants) | 2
  Week 3 Pre-dose | 4530 (53.7)
  Week 5 Pre-dose: number analyzed (Participants) | 2
  Week 5 Pre-dose | 3440 (62.9)
  Week 9 Pre-dose: number analyzed (Participants) | 1
  Week 9 Pre-dose | 5790 (NA) — Geometric Coefficient of Variation could not be calculated if the number of participants analyzed was less than 2.
  Week 13 Pre-dose: number analyzed (Participants) | 1
  Week 13 Pre-dose | 6360 (NA) — Geometric Coefficient of Variation could not be calculated if the number of participants analyzed was less than 2.
  Week 17 Pre-dose: number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant regardless of its causal relationship to study treatment. An AE can be any unfavorable and unintended sign (including any clinically significant abnormal laboratory test result), symptom, or disease temporally associated with the use of the study drug, whether or not it was considered to be study drug related.
Time Frame: Up to approximately 76 months
Population: The analysis population consisted of all allocated participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-3795
Number analyzed (Participants) | 4
Participants | 4

12. Secondary Outcome: Number of Participants Who Discontinued Study Intervention Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant regardless of its causal relationship to study treatment. An AE can be any unfavorable and unintended sign (including any clinically significant abnormal laboratory test result), symptom, or disease temporally associated with the use of the study drug, whether or not it is considered to be study drug related.
Time Frame: Up to approximately 74 months
Population: The analysis population consisted of all allocated participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-3795
Number analyzed (Participants) | 4
Participants | 2

ADVERSE EVENTS:
Time Frame: Up to approximately 76 months
Description: Serious and Other adverse events (AEs) included all participants who received ≥1 dose of study drug. All-Cause Mortality included all allocated participants. Data are reported by treatment received.
Arm/Group | MK-3795
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3795 (N=4)
Aphasia (Nervous system disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3795 (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2)
Dry eye (Eye disorders) | 3 (3)
Photopsia (Eye disorders) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (3)
Vitreous floaters (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 4 (4)
Oral pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Herpes zoster cutaneous disseminated (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Mammogram abnormal (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Aphasia (Nervous system disorders) | 3 (4)
Cognitive disorder (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (6)
Neuralgia (Nervous system disorders) | 1 (2)
Post herpetic neuralgia (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3)
Irritability (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Macule (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor reserves the right to review all planned communications and manuscripts based on the results of this study. This reservation of right is not intended to restrict or hinder publication of any dissemination of study results, but to allow the Sponsor to confirm the accuracy of the data, to protect proprietary information, and to provide comments based on information that may not yet be available to the study Investigators.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT03108066/Prot_SAP_000.pdf